CLINICAL TRIAL: NCT03314636
Title: KRd Consolidation in Myeloma Patients With a Positive PET-CT After Standard First Line Treatment. A Phase II Study
Brief Title: Intensified Treatment With Carfilzomib in Myeloma Patients Still PET-positive After First Line Treatment.
Acronym: CONPET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Nordic Myeloma Study Group (Other)
Responsible Party: Principal Investigator, Fredrik Hellem Schjesvold, Head of Oslo Myeloma Center, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMSG25/16
Record Dates: First submitted 2017-09-08; First posted 2017-10-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-03

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — carfilzomib; Lenalidomide; Positron Emission Tomography Computed Tomography; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET-CT-positive patients (Experimental): Carfilzomib 20/36mg/m2 days 1,2,8,9,15,16 Lenalidomide 25mg days 1-21 Dexamethasone 40mg days 1,8,15,22 28 day cycles 4 cycles
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Device: PET-CT; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — See in arm description
Drug: Lenalidomide — See in arm description
Device: PET-CT — See in arm description
Drug: Dexamethasone — See in arm description

SUMMARY:
A PET-CT will be performed on patients with myeloma after a standard first-line treatment. The PET-positive patients will receive 4 cycles of Carfilzomb-Revlimid-Dexamethason (KRd), before a new PET-CT will be performed.

DETAILED DESCRIPTION:
Patients will be evaluated for inclusion after finishing first-line therapy, or after a sufficient amount of treatment in first-line, and a sufficient respons (VGPR). Eligible performed regimens are defined in the protocol. All patients will perform a PET-CT, and PET-negative patients will be excluded from protocol treatment. The PET-positive patients will do a minimal residual disease (MRD-)evaluation in the bone marrow before entering treatment. After 4 28day cycles of Carfilzomib-Revlimid-Dexamethason, a new MRD and a new PET-CT will be performed, as measures of outcome. Patients will continue treatment as written in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Prior confirmed diagnosis of multiple myeloma (2014).
2. Received standard first line treatment with at least partial response. Standard first line treatment is defined as

   * VRD, VTD or VCD followed by ASCT, or
   * MPV at least 6 cycles, or no further reduction in monoclonal component the last 2 cycles, or
   * Rd at least 9 cycles or no further reduction in monoclonal component the last 2 cycles.
3. Carfilzomib naïve.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. Absolute neutrophil count (ANC) ≥ 0,5 x 109/L) and platelet count >35 x 109/L.
6. At least very good partial remission (VGPR) from first line treatment

Exclusion Criteria:

1. Change of first line treatment because of stabile or progressive disease.
2. Major surgery within 28 days before enrollment.
3. Radiotherapy within 14 days before enrollment, but if the involved field is small, 7 days will be considered a sufficient interval before onset of the treatment.
4. Glucocorticoid therapy within the 14 days prior to inclusion that exceeds a cumulative dose of 160 mg dexamethasone or 1000 mg prednisone.
5. Central nervous system involvement.
6. Uncontrolled heart disease, including congestive heart failure (NYHA III-IV), uncontrolled angina pectoris, uncontrolled conduction abnormalities, acute diffuse infiltrative pulmonary disease, pericardial disease or myocardial infarction within 6 months prior to enrollment
7. Uncontrolled hypertension or uncontrolled diabetes despite medication
8. Active hepatitis B or C infection or known human immunodeficiency virus (HIV) positivity.
9. Another active malignancy. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
10. Primary plasma cell leukemia, systemic AL amyloidosis, Waldenströms macroglobulinemia, POEMS syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
PET negativity after induction | 1 month after induction
  How many of PET positive patients will become PET negative after treatment

SECONDARY OUTCOMES:
PET correlation with MRD Euroflow | 1 month after induction
  Before intervention all patients are PET-CT positive. The investigators will measure minimal residual disease (MRD) with immuno-flow cytometry, at the same timepoint, and describe how many of the PET-CT patients, are MRD-negative and how many are MRD-positive. After the intervention the investigators will again do PET-CT and MRD by flow cytometry. The investigators will then describe how many PET-positive patients are MRD-positive and how many are MRD-negative. As well, the investigators will describe the same in the PET-CT negative patients.

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (2):
  - Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Oslo University Hospital, Oslo, Norway
- Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenberg T, Moller S, Abildgaard N, Norgaard JN, Lysen A, Tsykonova G, Joao C, Vangsted A, Schjesvold F, Nielsen LK. Health-Related Quality of Life During Carfilzomib-Lenalidomide-Dexamethasone Consolidation: Findings From the Multiple Myeloma CONPET Study. Eur J Haematol. 2025 Mar;114(3):517-527. doi: 10.1111/ejh.14358. Epub 2024 Dec 5. PMID 39638553